CLINICAL TRIAL: NCT03695341
Title: Fulvestrant Versus Everolimus Plus Exemestane for Patients With Metastatic Breast Cancer Resistant to Aromatase Inhibitors: the Clinical Experience From Real -World
Brief Title: 500mg Fulvestrant Versus Everolimus Plus Exemestane in MBC Patients Refractory to Previous AI
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-3
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: Endocrine Therapy; Fulvestrant; Everolimus
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fulvestrant: Fulvestrant 500mg per month (D1, D28, q28d), with a loading dose 500mg of first dose at D15
- Everolimus plus Exemestane: Everolimys 10 mg or 5 mg daily; Exemestane 25mg per day

SUMMARY:
500mg Fulvestrant versus Everolimus plus Exemestane in MBC patients refractory to previous AI

DETAILED DESCRIPTION:
Fulvestrant versus Everolimus plus Exemestane for patients with Metastatic Breast Cancer resistant to Aromatase Inhibitors: the clinical experience from real -world

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with ER/PR+，HER2- Metastatic Breast Cancer
2. Patients who were refractory to previous Aromatase Inhibitors
3. Patients treated with Fulvestrant or Everolimus plus Exemestane in any line in metastatic setting in Fudan University Shanghai Cancer Center，starting from 2013.06.01-2016.06.01
4. Available medical history

Exclusion Criteria:

1.Incomplete medical history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Xie Y, Gong C, Zhao Y, Zhang J, Zhang S, Wang L, Chen S, Hu X, Wang B. Comparative Treatment Patterns and Outcomes of Fulvestrant versus Everolimus Plus Exemestane for Postmenopausal Metastatic Breast Cancer Resistant to Aromatase Inhibitors in Real-World Experience. Ther Clin Risk Manag. 2020 Jun 30;16:607-615. doi: 10.2147/TCRM.S255365. eCollection 2020. PMID 32636632